CLINICAL TRIAL: NCT03740516
Title: Expanded Access for CC-10004
Status: No longer available | Type: Expanded Access
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-10004
Record Dates: First submitted 2018-10-31; First posted 2018-11-14 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Bechet's Disease
Keywords: Expanded Access; Compassionate Use
MeSH Terms: interventions — apremilast

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: CC-10004 — CC-10004 will be administered orally
  Other Names: Apremilast, Otezla

SUMMARY:
This is an expanded access program (EAP) for eligible participants designed to provide access to CC-10004.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Celgene, Summit, New Jersey, United States